CLINICAL TRIAL: NCT06837038
Title: Clinical Study of Rhythmic Auditory Stimulation for Gait Disorders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: YiCheng Zhu (Other)
Responsible Party: Sponsor-Investigator, YiCheng Zhu, Project Leader, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K7442; 2022-PUMCH-D-007 (Other Grant/Funding Number: Clinical research program of the central high-level hospital)
Record Dates: First submitted 2025-02-05; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-12

CONDITIONS: Hemiplegia Due to Stroke; Parkinson Disease; Parkinsonian Syndrome
Keywords: Rhythmic auditory stimulation; Hemiplegia after stroke; Parkinsonism syndrome; Gait disorders; Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rhythm intervention group (Experimental)
  Interventions: Device: rhythmic auditory stimulation
- Active control group (Sham Comparator)
  Interventions: Device: No rhythm stimulation

INTERVENTIONS:
Device: rhythmic auditory stimulation — The intervention group was treated with a gait rhythm device under the supervision of the researchers. The complete gait training was conducted once a day for 15 minutes for 7 consecutive days. Each patient wore inertial sensors at both ankles during gait training to collect gait information during walking.
  Arms: Rhythm intervention group
Device: No rhythm stimulation — The control group received gait training without rhythmic auditory stimulation under the supervision of the researchers. The complete gait training was conducted once a day for 15 to 20 minutes for 7 consecutive days. Each patient wore inertial sensors at both ankles during gait training to collect gait information during walking.
  Arms: Active control group

SUMMARY:
The aim of this clinical trial was to determine whether rhythmic auditory stimulation is effective in treating gait disorders in patients with post-stroke hemiplegia, primary Parkinson's disease, and various parkinsonism syndromes. The main questions it aims to answer are:

Does rhythmic auditory stimulation increase walking speed in patients with gait disorders? To determine whether rhythmic auditory stimulation is effective in treating gait disorders, researchers will compare a gait rhythmometer with an active control that does not receive rhythmic stimulation.

Participants will:

Gait training was conducted once a day for 15 minutes for 7 consecutive days Resting-state functional magnetic resonance imaging (fmri) was performed before and after treatment Feedback on subjective improvement at the end of the 7-day treatment

ELIGIBILITY:
For post-stroke hemiplegia

Inclusion criteria :

* Age 50-80 years old
* One or more strokes (cerebral infarction or cerebral hemorrhage), with the most recent stroke occurring at least 6 months earlier
* Walking independently without a cane or walking aid with obvious gait asymmetry
* 0.4m/s< baseline velocity <0.8m/s
* Sufficient hearing, vision and comprehension to complete motor function tests
* Patients were willing and able to participate in all study procedures and signed informed consent
* No other rehabilitation treatment was received at present

Exclusion Criteria:

* Unable to cooperate with the motor function test
* Uncontrolled hypertension
* Myocardial infarction within the past 3 months
* With bone and joint diseases, such as a history of lower limb fracture within 1 year, waist and lower limb bone and joint surgery, bone and joint deformity seriously affecting walking, etc.
* Except for stroke, there was no parkinsonism, myasthenia gravis, poliomyelitis and other nervous system diseases affecting the walking function of patients.

For primary Parkinson's disease (PD)

Inclusion criteria:

* Age 50-80 years old
* PD met the diagnostic criteria of Chinese Diagnostic Criteria for Parkinson's Disease (2016 edition)
* Obvious panic gait, freezing gait or slow gait, but can walk independently without the use of a cane or walking aid
* Hoehn-Yahr (H-Y) stage 2-4
* 0.4m/s< baseline velocity <0.8m/s
* Sufficient hearing, vision and comprehension to complete motor function tests
* Patients were willing and able to participate in all study procedures and signed informed consent
* No other rehabilitation treatment was received at present

Exclusion criteria:

* Unable to cooperate with the motor function test
* Uncontrolled hypertension
* Myocardial infarction within the past 3 months
* With bone and joint diseases, such as a history of lower limb fracture within 1 year, waist and lower limb bone and joint surgery, bone and joint deformity seriously affecting walking, etc
* There was no stroke, myasthenia gravis, poliomyelitis and other neurological diseases affecting the walking function except for primary Parkinson's disease

For Parkinsonism syndrome:

Inclusion criteria:

* Age 50-80 years old
* All parkinsonism syndrome except primary Parkinson's disease, including but not limited to drug-induced parkinsonism, multiple system atrophy, cerebral small vessel disease-related parkinsonism, etc
* obvious panic gait, freezing gait or slow gait, but can walk independently without the use of a cane or walking aid
* 0.4m/s< baseline velocity <0.8m/s
* Sufficient hearing, vision and comprehension to complete motor function tests
* Be willing and able to participate in all study procedures and sign informed consent
* No other rehabilitation treatment was received at present.

Exclusion criteria:

* Unable to cooperate with the motor function test
* Uncontrolled hypertension
* Myocardial infarction within the past 3 months
* With bone and joint diseases, such as a history of lower limb fracture within 1 year, waist and lower limb bone and joint surgery, bone and joint deformity seriously affecting walking, etc
* There was no stroke, myasthenia gravis, poliomyelitis and other neurological diseases that affected the walking function except for parkinsonism

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | 10 days
  The difference between the gait speed measured on the third day after the completion of the seven gait sessions and the baseline gait speed

SECONDARY OUTCOMES:
Stride length | 10 days
  The difference between the stride length (left and right) measured on the third day after the completion of the seven gait sessions and the baseline stride length.
Stride frequency | 10 days
  The difference between the stride frequency (left and right) measured on the third day after the completion of the seven gait sessions and the baseline stride frequency.
Stride speed | 10 days
  The difference between the stride speed (left and right) measured on the third day after the completion of the seven gait sessions and the baseline stride speed.
Swing speed | 10 days
  The difference between the swing speed (left and right) measured on the third day after the completion of the seven gait sessions and the baseline swing speed.
Standing phase | 10 days
  The difference between the standing phase (left and right) measured on the third day after the completion of the seven gait sessions and the baseline standing phase.
Turn time | 10 days
  The difference between the turn time measured on the third day after the completion of the seven gait sessions and the baseline turn time.
Patient's SUBJECTIVE assessment | 10 days
  All subjects were asked about their subjective feelings using a uniform questionnaire, including the following questions: Did the patient's gait problems improve after 7 days of treatment? If there has been improvement, in what ways? (Step speed, stride length, symmetry, turn time, etc.)
Resting-state functional magnetic resonance imaging | 10 days
  At baseline and on the third day after completion of the 7-day gait treatment, 3T resting-state functional magnetic resonance imaging (rs-fMRI) was performed to compare the changes of local neural activity, including amplitude of low frequency fluctuation (ALFF) and functional connectivity density (FCD).

CONTACTS AND LOCATIONS:
Overall Officials: Yicheng Zhu, Study Director
Locations (1):
- Department of Neurology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China